CLINICAL TRIAL: NCT05852392
Title: Parent-focused Redesign for Encounters, Newborns to Toddlers (PARENT) Trial: Comparing Two Models of Well-Child Care for Black Families
Brief Title: Comparing Two Models of Well-Child Care for Black Families
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Nationwide Children's Hospital (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Tumaini Coker, Division Chief, General Pediatrics, Seattle Children's Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00004147
Record Dates: First submitted 2023-04-13; First posted 2023-05-10 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Pediatric; Well Child Care
Keywords: Community Health Workers; Well Child Care; Black Children; Black Families; Preventive Care; Early Childhood; Patient-centered economic outcomes

STUDY DESIGN:
Intervention Model Description: We will use a stepped wedge design, in which each of 12 clinical practice site starts in the control group, and then sequentially (by random assignment) moves to become intervention. Under "enrollment" below, we list the number of clinics to be randomized, as individual participants are not randomized or enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted PARENT Model (Experimental): PARENT is a team-based approach to care that utilizes a community health worker (called a "coach") as part of the WCC team to provide comprehensive and family-centered preventive care services, address concerns related to family social needs, and decrease reliance on the clinician as the sole provider of preventive care services. The coach independently meets with the family at every early childhood well-child care visit to provide anticipatory guidance, social needs screening, developmental screening, and connection to needed community resources. All NCH-PCN practices will start in the control group, and then sequentially (by random assignment) move to become intervention. Practices will implement the adapted PARENT model for all well-visits, newborn through 15 months of age, and have a 9-month implementation exposure period to ensure that children ≤15 months of age at the practice have received the intervention; thereafter the practices maintain the intervention.
  Interventions: Other: Adapted PARENT Model
- Traditional Well-Child Care (No Intervention): Our comparator is traditional well-child care, which follows national preventive care guidelines including structured and standardized developmental and social needs screening, and is in widespread use. These are well-child care visits led by the primary care clinician without a community health worker. All NCH-PCN practices will start in the control group, and then sequentially (by random assignment) move to become intervention.

INTERVENTIONS:
Other: Adapted PARENT Model — PARENT is a team-based approach to care that utilizes a clinic-based community health worker as part of the WCC team to provide comprehensive and family-centered preventive care services.
  Arms: Adapted PARENT Model

SUMMARY:
Parent-focused Redesign for Encounters, Newborns to Toddlers (PARENT) is a team-based approach to care that utilizes a community health worker in a health educator role ("Parent's Coach") to provide many of the Well-Child Care (WCC) services that children and families should receive, addresses specific needs faced by families in low-income communities, and decreases reliance on the clinician as the primary provider of WCC services. The model was developed in partnership with clinics and parents in low-income communities and previously tested among largely Latino, Medicaid-insured populations. The aims of this study are to (1) Adapt the PARENT intervention to meet the needs of a diverse, largely Black population of underserved families, (2) Determine the effect of adapted PARENT on receipt of nationally recommended preventive care services, emergency department utilization, and parent experiences of care, (3) Determine whether the effectiveness of adapted PARENT differs by family-level factors, (4) Explore parents' experiences in receiving adapted PARENT, (5) Examine the economic impact of adapted PARENT from the parent stakeholder perspective, (6) Examine the economic impact of adapted PARENT from the pediatric provider and clinic stakeholder perspective, and (7) Examine the economic impact of adapted PARENT on healthcare utilization, from the perspectives of parents and families.

This study will evaluate the effectiveness of the adapted PARENT model as compared to traditional guideline-based WCC and assess the patient-centered economic outcomes of the adapted PARENT model.

DETAILED DESCRIPTION:
Clinical Practice Redesign can lead to innovative systems that improve preventive care for racial and ethnic minority children in low-income communities. Although several strategies to redesign the structure of Well-Child Care (WCC) have been proposed and studied, there are few evidence-based comprehensive models that are financially sustainable alternatives to current WCC. The Parent Focused Redesign for Encounters, Infants to Toddlers (PARENT) is a comprehensive early childhood WCC delivery model designed to improve the delivery of WCC for infants and toddlers in low-income communities. PARENT includes a community health worker as part of a team-based approach to WCC. The "Parent's Coach" partners with the clinician to independently provide comprehensive and family-centered care that includes anticipatory guidance, social needs screening, developmental screening, and connection to needed community resources. The Parent's Coach reduces the reliance on a clinician as the sole primary provider of routine WCC services. The intervention changes the structure of WCC by adding the Parent's Coach to the team (personnel), and changing the process, or provision of care, which impacts the receipt of preventive care, and thus health outcomes.

In previous trials of PARENT, among a predominately Latino population of Medicaid-insured children, we have reported intervention effects of better parent experiences of care, greater receipt of preventive care services, and more effective utilization of care. Although these trials were not powered for sub-analyses by race, exploratory analyses indicate that while Black and Latino families had similar intervention effects for receipt of services, Black families did not have the positive intervention effects on parent experiences of care or the reduction of emergency department (ED) visits that Latino families did. Thus, adaptation, implementation, and testing of PARENT in a trial with a large sample of Black families is needed to optimize outcomes for Black families. PARENT will be adapted, implemented, and tested in clinics that serve a large proportion of low-income Black families, providing findings to aid our understanding of how the intervention can be adapted to meet the needs of low-income Black families.

The adapted intervention, if found to be more effective than usual care in providing family-centered, comprehensive preventive care services to families, has the potential to be implemented and disseminated to other clinical settings that serve a large proportion of children in low-income areas. However, our stakeholders for early childhood WCC will require additional information on family-centered economic outcomes to make decisions regarding the implementation and dissemination of this new model for early childhood preventive care. To address this need, we will examine patient-centered economic outcomes during the stepped wedge trial of the adapted intervention that will provide additional information to help WCC stakeholders make decisions about the delivery of care for early childhood WCC services.

The study team will collaborate with investigators at Nationwide Children's Hospital Primary Care Network (NCH-PCN) to conduct this study. NCH-PCN is one of the largest Children's Hospital owned primary care networks in the country. Its 12 practices serve a patient population that is over 96% publicly insured, 50% Black, and 16% Latino. Collaboration on this study represents a unique opportunity to meet a clinical need at NCH-PCN and address key research questions of PARENT adaptation, implementation, and impact for Black families.

The study will conducted using a stepped wedge randomized trial design in order to evaluate the intervention's effectiveness as well as its patient-centered economic outcomes.

ELIGIBILITY:
Inclusion Criteria:

Participants are not individually recruited or enrolled; rather we collect de-identified Electronic Health Record (EHR) and administrative data on all children in the practices who:

1. are age ≥9 and ≤15 months on day of data collection,
2. have ≥1 visit at the practice in previous 9 months
3. are insured by Partners for Kids, the Accountable Care Organization (ACO) for NCH-PCN

Exclusion Criteria:

* N/A

Ages: 9 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Receipt of preventive care services | Every 9 months, up to 5 years
  Child and parent receipt of three key preventive care services: anticipatory guidance, social needs screening, and structured developmental screening
Healthcare Utilization | Every 9 months, up to 5 years
  Emergency department visits
Parent Experiences of Care | Every 9 months, up to 5 years
  Family-Centeredness Measure

SECONDARY OUTCOMES:
Receipt of additional preventive care services | Every 9 months, up to 5 years
  Receipt of a) social needs referral (e.g., to a food bank), b) successful connection with social needs source (e.g., parent reports accessing food bank), c) developmental or behavioral referral (e.g., Early Intervention Center), and d) successful connection with developmental needs source (e.g., visit at Early Intervention completed).
Other Healthcare Utilization | Every 9 months, up to 5 years
  WCC and acute care visits, and hospitalizations
"At-risk" for developmental delay | Every 9 months, up to 5 years
  Identified as "at-risk" following developmental screening

OTHER OUTCOMES:
Provider-parent visit time | Every 9 months, up to 5 years
  Time stamped number of minutes that provider spent in visit with family
Coach-parent visit time | Every 9 months, up to 5 years
  Time stamped number of minutes that coach spent in visit with family
Registered Nurse/Medical Assistant (RN/MA)-parent visit time | Every 9 months, up to 5 years
  Time stamped number of minutes that the Registered (RN) or Medical Assistant (MA) spent in visit with family
Total visit time | Every 9 months, up to 5 years
  Time stamped number of minutes family spent at visit (from check in to discharge)
Provider documentation time | Every 9 months, up to 5 years
  Time stamped number of total minutes that provider spent in EHR in the visit encounter form (from opening of encounter form to closing/signing it).

CONTACTS AND LOCATIONS:
Overall Officials: Tumaini Coker, MD, MBA, Principal Investigator — Seattle Children's Hospital
Locations (2):
- United States (2):
  - Nationwide Children's Hospital, Columbus, Ohio
  - Seattle Children's Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Patient-Centered Outcomes Research Institute (PCORI): Comparing Two Models of Well-Child Care for Black Families — https://www.pcori.org/research-results/2022/comparing-two-models-well-child-care-black-families